# STATISTICAL ANALYSIS PLAN

# **Mi-ECMO Study**

NCT02940327

A FEASIBILITY STUDY TO CONSIDER THE RELATIONSHIP BETWEEN MARKERS OF RED CELL DAMAGE, INFLAMMATION AND THE RECOVERY PROCESS OF NEWBORNS REQUIRING EXTRACORPOREAL MEMBRANE OXYGENATION (ECMO) FOR PERSISTENT PULMONARY **HYPERTENSION OF THE NEWBORN (PPHN)** 

**SAP Version:** 1.0

Date: 01-May-2018

**Based on protocol** 

Protocol number: **UNOLE 0553** 

Version: 4.0

27-Feb-2017 Date:

Sponsor Name: University of Leicester Sponsor Address: Research Support Office

> **University Road** Leicester, LE1 7RH

Study Statistician: Florence Lai

University of Leicester Glenfield Hospital Leicester, LE3 9QP

Chief Investigators: Mr Gavin Murphy

**Professor of Cardiac Surgery** University of Leicester Glenfield Hospital Leicester LE3 9QP

Dr Simon Robinson

Paediatric Intensivist and ECMO Consultant

Glenfield Hospital Leicester LE3 9QP













# Contents

| Glossa | ry / abbreviations | 3 |
|--------|-----------------------------------------|----|
| 1. In | ntroduction | 4 |
| 1.1 | Aims and Objectives | 4 |
| 1.2 | Study Design | 5 |
| 1.3 | Sample Size | 5 |
| 1.4 | Study population | 5 |
| In | nclusion Criteria | 5 |
| Ex | xclusion criteria | 6 |
| 1.5 | Schedule of Major Assessments | 6 |
| 2. Er | ndpoints | 7 |
| 2.1 | Primary outcomes | 7 |
| 2.2 | Secondary outcomes | 7 |
| 2.3 | Target conditions | 8 |
| 3. Aı | nalysis Sets/Populations | 9 |
| 3.1 | Full analysis set population | 9 |
| 3.2 | Safety population | 9 |
| 3.3 | Protocol deviations | 9 |
| 4. St | tatistical Methodology | 9 |
| 4.1 | Timing of Analysis and Interim Analysis | 9 |
| 4.2 | Disposition of Patients | 9 |
| 4.3 | Descriptive Analysis | 9 |
| 4.4 | Statistical Methods | 9 |
| 4.5 | Subgroup analysis | 10 |
| 4.6 | Multiple Comparisons | 10 |
| 4.7 | Handling of Missing Data | 10 |
| 5. Sa | afety Analysis | 10 |
| 5.1 | Adverse events reporting | 10 |
| 5.2 | Expected adverse events | 10 |
| 6. Re | eferences | 11 |
| Appen | dix A List of variables for reporting | 12 |

# Glossary / abbreviations

AE Adverse event
AKI Acute kidney injury

ARG1 Arginase 1

CD Cluster of differentiation

CDH Congenital diaphragmatic hernia

CO₂ Carbon dioxide CmH₂O Centimetre of water CPB Cardiopulmonary bypass

CRF Case report form

CRRT Continuous renal replacement therapy
CSCTT Cardiac surgery clinical trials team
ECMO Extra-corporeal membrane oxygenation

EDTA Ethylenediaminetetraacetic acid FACS Fluorescence activated cell sorting

FiO<sub>2</sub> Fraction of inspired oxygen GFR Glomerular filtration rate

Hb Haemoglobin

HFOV High frequency oscillatory ventilation

HMOX1 Heme oxygenase 1 ICU Intensive care unit

ICAM Intercellular adhesion molecule

IL Interleukin

INOS Inducible nitric oxide synthase

KDIGO The International Society of Nephrology: Kidney Diseases Improving Global

Outcomes (KDIGO) definition of acute kidney injury (AKI)

MAS Meconium aspiration syndrome
MABP Mean arterial blood pressure
MCP Monocyte chemoattractant protein

MI Myocardial infarction

MP Microparticles MV Microvesicles

NGAL Neutrophil gelatinase associated lipocalin

NO Nitric oxide

pCO<sub>2</sub> Partial pressure of carbon dioxide
 PEEP Positive End Expiratory Pressure
 PICU Paediatric intensive care unit
 PIL Patient information leaflet

PPHN Persistent pulmonary hypertension of the newborn

RDS Respiratory distress syndrome

SaO<sub>2</sub> Oxygen saturation

SIRS Systemic inflammatory response syndrome

SOP Standard operating procedures TNF-α Tumour necrosis factor – alpha

#### 1. Introduction

The Mi-ECMO study is a pilot feasibility study to consider the relationship between markers of red cell damage, inflammation and the recovery process of newborns requiring Extra-Corporeal Membrane Oxygenation (ECMO) for Persistent Pulmonary Hypertension of the Newborn (PPHN).

This Statistical Analysis Plan (SAP) describes the analysis and reporting for the Mi-ECMO study. It outlines the planned analysis to be performed on the data. Exploratory post-hoc or unplanned analysis not necessarily identified in this SAP may be performed as required.

#### 1.1 Aims and Objectives

#### **Hypothesis**

The primary hypothesis is that damage to red blood cells by the exposure to the ECMO circuit will result in inflammatory responses that mitigate against successful weaning from ECMO for PPHN.

The secondary hypothesis are:

- 1. Damage to red cells will result in platelet, leukocyte and endothelial activation.
- 2. Markers of platelet, endothelial and leukocyte activation are indicators of lung inflammation and injury severity and hence lung recovery.
- 3. Markers of platelet, endothelial and leukocyte activation are indicators of kidney injury severity and hence acute kidney injury.
- 4. Granulocyte and platelets activation are secondary to rising redox potential and the levels of activation will correlate with longer intubation times and more severe organ injury.
- 5. Markers of platelet, endothelial and leukocyte activation have diagnostic and prognostic utility for the prediction of key clinical events including delayed time to recovery, acute kidney injury in paediatric patients undergoing ECMO for PPHN.

## **Objectives**

The Mi-ECMO study was designed to be a feasibility study, and the results will be used to assist with the design of a prospective observational study that will test the above hypotheses. The objectives of the study are:

- 1. To determine the recruitment rates and patient flows for 24 patients recruited for the feasibility study.
- 2. To determine the withdrawal rate and the completeness of follow-up and data collection in a paediatric population at high risk for death and major morbidity.
- 3. To collect data on primary and secondary outcomes of interest, which may be used to model the sample sizes and outcomes in future study.
- 4. To collect data on perception of family members, whose children participate in the study, as to their understanding of the screening and consent process (Appendix 1).

### Changes in hypothesis

Due to the lack of ethnical approval, this study is not conducting analysis of bronchial aspirates, and measuring markers of oxidative stress and MV levels. The following secondary hypothesis which were stated in the study protocol have not been included in this SAP:

- 1. The level of oxidative stress will correlate with type shifts in pulmonary macrophages, tissue iron deposition and organ injury.
- 2. Ability to raise anti-oxidative response, measured by Heme Oxigenase-1 (HMOX 1) expression, will correlate with shorter intubation times and less severe kidney and lung injury.
- 3. Markers of anti-oxidative response and oxidative stress levels have diagnostic and prognostic utility for the prediction of key clinical events including delayed time to recovery, acute kidney injury in paediatric patients undergoing ECMO for PPHN.

Correspondingly, all related secondary outcomes would not be included in this SAP.

# 1.2 Study Design

The Mi-ECMO study is a prospective, single-centre observational feasibility study.

#### 1.3 Sample Size

The Mi-ECMO study enrolled 24 patients. There was not a formal power calculation for this feasibility study. The sample size was based on the observations from a similar study, p-MiVAKI which had recruited 24 paediatric patients and was able to demonstrate differences in the primary outcomes, markers of platelets, leukocyte and endothelial activation, between those who did and did not develop AKI, and between those did and did not receive transfusion.

# 1.4 Study population

The study was conducted at Glenfield Hospital, a regional ECMO centre in the UK, the University Hospitals of Leicester NHS Trust. The Glenfield Hospital is a national paediatric referral centre and provides ECMO support across UK from phone consultation to onsite cannulation and transport on ECMO. This unit performs over 60 neonatal and paediatric ECMO per year, of which at least 40 are expected to be performed for the treatment of PPHN in infants.

Participants of this study were consecutive patients referred to the Glenfield Hospital according to the ECMO referral system who match the following study criteria.

#### Inclusion Criteria

Participant may enter study if all of the following apply:

- 1. Patients with a diagnosis of PPHN
- 2. Patients that require ECMO support as determined by the ECMO team
- 3. Patients aged less than 30 days
- 4. Emergency consent obtained within 12 hours from cannulation, and ultimately full consent

# Exclusion criteria

Participant may not enter study if any of the following apply:

- 1. PPHN is caused by a congenital heart pathology
- 2. ECMO is required for a congenital heart disease
- 3. Lack of consent

# 1.5 Schedule of Major Assessments

| | Baseline<br>(12h after<br>ECMO start<br>+/- 6 hrs) | Day 1<br>(24 hrs<br>+/- 12 hrs) | Day 2<br>(48h<br>+/- 12 hrs) | Day 3<br>(72h +/-<br>12 hrs) | 24h after<br>decannulation/<br>prior to ECMO stop for<br>death or withdrawal<br>(+/- 12 hrs) |
|---|---|---|---|---|---|
| Eligibility | ✓ | | | | |
| Written emergency consent | <b>✓</b> | | | | |
| Trial Registration | ✓ | | | | |
| Clinical outcomes | ✓ | ✓ | ✓ | <b>✓</b> | ✓ |
| Serious adverse event monitoring | <b>✓</b> | ✓ | ✓ | <b>√</b> | ✓ |
| Bloods: Full blood<br>count | ✓ | ✓ | ✓ | ✓ | ✓ |
| Bloods: Cytokines, total iron, non-transferrin-bound iron | ~ | <b>✓</b> | <b>~</b> | ~ | <b>√</b> |
| Bloods: Platelets and leukocyte activation | ✓ | ✓ | ✓ | <b>✓</b> | ✓ |
| Bloods: MV analysis | ✓ | ✓ | ✓ | ✓ | ✓ |
| Respiratory Sample:<br>ferrocyanide, oxidative<br>stress | 1 | <b>✓</b> | <b>√</b> | <b>✓</b> | <b>√</b> |
| Urine sample & volume: NGAL | ✓ | ✓ | ✓ | ✓ | ✓ |
| Questionnaire on perception of family members | | | | | <b>√</b> |

## 2. Endpoints

A list of variables to be evaluated and reported in the statistical analysis is provided in the Appendix.

## 2.1 Primary outcomes

Markers of cellular activation including platelet, leukocyte and endothelial cell activation in arterial blood at baseline (12 hours after ECMO commencement) and then at 24, 48 and 72 hours post commencement and at weaning (24 hours after decannulation) or immediately prior to ECMO support being stopped in case of death or treatment withdrawal.

Markers of cellular activation include CD41, PAC-1 and CD62P for platelets, CD64 and CD163 for leukocytes, CD14, CD16, and CD41 for platelet-leukocyte aggregates, as well as circulating ICAM and E-selectin for endothelial injury.

# 2.2 Secondary outcomes

#### Clinical outcomes

- 1. Serum haemoglobin levels.
- 2. Time to wean from ECMO.
- 3. Percentage of patients weaned from ECMO within 7 days
- 4. AKI as defined by the KDIGO pediatric definition (Table 1)
- 5. AKI as defined based on the neonatal modification (Table 2)
- 6. Heart injury as determined by serum troponin levels.
- 7. Renal inflammation as determined by urine NGAL concentrations.
- 8. Allogenic red cell transfusion volume.
- 9. Non red cell transfusion volume.
- 10. Time to discharge from Glenfield Hospital ICU.
- 11. Time to Glenfield Hospital discharge.
- 12. Measures of haemoglobin metabolism e.g. serum hepcidin, serum haptoglobin, transferrin saturation, serum ferritin, plasma labile iron concentrations.
- 13. Inflammatory cytokines in serum, measured by IL-6, IL-8, TNFα, MCP-1 and MIP-1.
- 14. Other adverse events not specified above.

#### Feasibility outcomes

- 15. Recruitment, sampling rates, and Withdrawal rates
- 16. Protocol adherence including clinical and laboratory protocol adherence
- 17. Data completeness
- 18. Experience of parents/ family/ guardians in relation to the screening, consent and study procedures based on a questionnaire

**Table 1**. Pediatric KDIGO-staging system for acute kidney injury, as per reference [1], with modified Stage 3 as per the pRIFLE definition [2].

| Stage | Serum creatinine (SCr) criteria | Urine output criteria |
|---|---|---|
| 1 | SCr ≥ 26 μmol/L increase <u>or</u><br>SCr ≥1.5- to 2-fold from baseline | <0.5 ml/kg/hr for > 6 consecutive hrs |
| 2 | SCr ≥ 2 to 3-fold from baseline | <0.5 ml/kg/hr for > 12 hr |
| 3 | SCr ≥3-fold from baseline or<br>SCr ≥ 354 µmol/L or<br>Renal replacement therapy irrespective of stage or<br>*Decrease in estimated Creatinine Clearance (eCrCl) to less than<br>35 mL/min/1.73 m² using the Schwartz equation:<br>eCrCl(mL/min/1.73 m²) = (36.2 × Height in cm) / Creatinine in<br>µmol/L | <0.3 ml/kg/hr for > 24 hr<br>or anuria for 12 hr |

The above criteria include both an absolute and a relative change in creatinine to accommodate variations related to age, gender, and body mass index and to reduce the need for a baseline creatinine but do require at least two creatinine values within 48 hours. Only one criterion (creatinine or urine output) has to be fulfilled to qualify for a stage. 200% to 300% increase = 2- to 3-fold increase. Given wide variation in indications and timing of initiation of renal replacement therapy (RRT), individuals who receive RRT are considered to have met the criteria for stage 3 irrespective of the stage they are in at the time of RRT. The modified stage 3 criteria for children\* reflect the observation that infants with small body mass may be unable to generate high serum creatinine values.

**Table 2**. Neonatal acute kidney injury definition – modification from KDIGO pediatric AKI definition [3].

| Stage | Serum creatinine (SCr) criteria<br>Neonatal modification: 2015-2016 | Urine output criteria<br>Neonatal modification 2016 |
|---|---|---|
| 1 | SCr ≥ 26 μmol/L increase <u>or</u><br>SCr ≥1.5- to 2-fold from baseline | ≤1 ml/kg/hr for 24 hr |
| 2 | SCr ≥ 2 to 3-fold from baseline | ≤0.5 ml/kg/hr for 24 hr |
| 3 | SCr ≥3-fold from baseline <u>or</u><br>SCr ≥ 221 µmol/L <u>or</u><br>Renal replacement therapy irrespective of stage | ≤0.3 ml/kg/hr for 24 hr |

#### 2.3 Target conditions

- Prolonged ECMO defined as patients remained on ECMO at day 7 (duration of ECMO >168 hours)
- 2. AKI as defined by the KDIGO stage 1, 2 or 3 using the paediatric AKI definition (Table 1).
- 3. AKI as defined by the KDIGO stage 1, 2 or 3 using the serum creatinine criteria for the neonatal AKI definition (Table 2).

# 3. Analysis Sets/Populations

# 3.1 Full analysis set population

The full analysis set population comprises all recruited patients with full consent. This population comprises 24 patients. All analyses of clinical outcomes will be carried out on the full analysis set population.

#### 3.2 Safety population

The safety population comprises all recruited patients with either emergency consent or full consent even those withdrew from the study. This population will be used for safety analyses.

#### 3.3 Protocol deviations

Potential deviations from the protocol and their categorisation into major/minor are to be discussed by the trial team. In general, protocol deviations would be considered as major if they could potentially lead to biased estimations of primary or secondary endpoints (e.g. entered into the study in error). Time window violations are generally not considered as major protocol deviations.

# 4. Statistical Methodology

# 4.1 Timing of Analysis and Interim Analysis

Analysis are to be performed when the final dataset with all laboratory data are ready. No interim analyse have been planned before the end of the recruitment phase.

#### 4.2 Disposition of Patients

Patient disposition will be presented with respect to recruitment rates, withdrawal rates, as well as protocol adherence including clinical and laboratory protocol adherence.

Data completeness will also be summarized.

#### 4.3 Descriptive Analysis

Descriptive analysis will be presented for demographic and baseline characteristics, as well as the primary and secondary outcomes, and targeted conditions described in Section 2. For categorical variables, numbers and percentages will be presented. For continuous variables, mean and standard deviation or median with lower and upper quartiles, as appropriate, will be presented.

#### 4.4 Statistical Methods

Mixed effects model with patient as random effect will be used to analyse outcomes measured at multiple time points. Logarithm transformation will be considered for skewed variables. Linear graphs showing the variation of the mean measurements over time will be displayed.

Exploratory analysis are to be carried out using mixed effects models to examine serial makers of cellular activation and their relationship with:

Duration on ECMO

- Transfusion volume
- Free cell haemoglobins
- NGAL concentrations
- Serum troponin levels
- Inflammatory cytokines

#### 4.5 Subgroup analysis

Exploratory analysis may be carried out to assess the relationship of cellular activation with the targeted subgroups:

- Patients on ECMO within 7 days vs 7+ days
- Patients with and without AKI

#### 4.6 Multiple Comparisons

There will be no adjustments for multiple comparisons, as this is a feasibility study to gather data on the primary and secondary outcomes for future study, and to explore the relationship between these outcomes to address the objectives described above.

#### 4.7 Handling of Missing Data

Lab measurements below the limit of quantification will be imputed as half the limit of quantification. Measurements above the limit of quantification will be imputed as the upper limit. No other missing values will be imputed.

#### 5. Safety Analysis

#### 5.1 Adverse events reporting

Data on adverse events are collected from ECMO commencement till hospital discharge. Adverse events shall be reported with the Safety Population.

### 5.2 Expected adverse events

The following adverse events are 'expected'.

- Suspected MI
- Cardiac arrest
- Heart or vessels perforation / chest opening
- Arrhythmias
- Pericardial effusion / cardiac tamponade
- Thromboembolic complications
- Haemodynamic support
- Pulmonary complications
- Renal complications
- Gastro-intestinal complications
- Neurological complications
- Bleeding
- Wound infection / infective complications (sepsis, septic shock etc)

Refer to the protocol for a full list of the expected adverse events.

# 6. References

- 1. KDIGO Clinical Practice Guideline for Acute Kidney Injury. Kidney Int Suppl, 2 (2012), pp. 122–123
- 2. Akcan-Arikan A, Zappitelli M, Loftis LL, Washburn KK, Jefferson LS, Goldstein SL. Modified RIFLE criteria in critically ill children with acute kidney injury. Kidney Int. 2007 May;71(10):1028-35. Epub 2007 Mar 28.
- 3. Zappitelli M, Ambalavanan N, Askenazi DJ, Moxey-Mims MM, Kimmel PL, Star RA, Abitbol CL, Brophy PD, Hidalgo G, Hanna M, Morgan CM, Raju TNK, Ray P, Reyes-Bou Z, Roushdi A, Goldstein SL. Developing a neonatal acute kidney injury research definition: a report from the NIDDK neonatal AKI workshop. Pediatr Res. 2017 Oct;82(4):569-573.

# Appendix List of variables for reporting

| Туре | Variable | Unit/Reference | Time points |
|---|---|---|---|
| Demographic, | Gestational age | week | |
| Characteristics | Preterm | Y/N | |
| at birth | Gender | M/F | |
| | Ethnicity | Caucasian /Other | |
| | Weight at birth | kg | |
| | Weight | kg | |
| | APGAR score at birth | 0 - 10 | |
| Clinical characteris | tics | | |
| Heart Rhythm | Sinus Rhythm | Sinus rhythm/AF /Heart block /Paced/Other | |
| Diagnosis | Diagnosis | Idiopathic PHN /MAS/CDH/ | |
| | - | pneumonia/RDS/PH/others | |
| Cardiac | LV function | mild / moderate / severe | |
| function | DV function | impairment | |
| function | RV function | mild / moderate / severe impairment | |
| | | None/Right to left/Left to right | |
| | Shunt | /Bidirectional | |
| | Shunt function | Restrictive / not restrictive | |
| Mechanical | Mechanical ventilation | Y/N | |
| ventilation | Modality | ., | |
| Cannulation | Haemodynamic instability | Y/N | prior to ECMO |
| | Blood priming | Y/N | p |
| | Clear priming | Y/N | |
| ECMO | MAP | mmHg | |
| Parameters | FiO2 on ECMO | % | Pre-ECMO (MAP |
| | FiO2 on ventilator | % | only); t=0, 12h, 24h, |
| | ACT | sec | 48h, 72h after start |
| | Pump flow | ml/min | of ECMO and before |
| | Sweep gas | ml/min | discontinuation |
| | RPM | revolutions/min | |
| Blood saving | Transexamic acid | Y/N | |
| J | Cell Saver (autologous) | Y/N | |
| Arrhythmia | Arrhythmia | -1 | |
| , | Cardioversion | Y/N | Placement, removal |
| | Defibrillation | Y/N | ECMO |

| Туре | Variable | Unit/Reference | Time points |
|---|---|---|---|
| Blood gas | рН | | |
| | pO2 | kPa | |
| | pCO2 | kPa | |
| | SaO2 | % | Pre-ECMP (PH, |
| | Hb | g/L | Lactate, PCO2, |
| | Glu | mmol/L | HCO3); t=0, 12h, |
| | Lactate | mmol/L | 24h, 48h, 72h after<br>start of ECMO and |
| | HCO3 | mmol/L | before |
| | Hct | % | discontinuation |
| | Na | mmol/L | |
| | K | mmol/L | |
| | Ca | mmol/L | |
| PICU | Lactates | mmol/L | t=0, 12, 24, 48 and |
| | PaO2/FiO2 | · | 72 hrs post PICU |
| | Total bilirubin | umol/L | admission & 24hrs |
| | Fibrinogen | g/L | after ECMO stop |
| | Urea | mmol/L | |
| | PIM2 score | Total Criteria Point Count | PICU admission |
| | PMODS score | Total Criteria Point Count | PICU admission & |
| | 1 10000 30010 | Total Criteria i Onic Count | 24h after ECMO stop |
| Medication | Inotrope Score | Total Criteria Point Count | |
| | Vasoactive-Inotrope score | Total Criteria Point Count | |
| Laboratory test | | | |
| Platelets, leukocyte | CD41, PAC-1, CD62P, CD64, | | |
| activation | CD163, CD14, CD16, CD41 | | |
| Granulocyte | CD11b | | <br>t=12h, 24h, 48h, 72h |
| Endothelial | ICAM, E-selectin | | ECMO, and 24h post |
| Cytokines | IL-6, IL-8, TNFα, MCP-1, MIP-1 | | ECMO and discharge |
| Iron | Total iron, non-transferrin-bour | nd iron | |
| Free Hb | Free cell Haemogloblins | 10 11011 | |
| Routine lab tests | Creatinine | umol/L | |
| | Adjusted Calcium | mmol/L | |
| | Alkaline Phosphatase | iu/L | |
| | ALT | iu/L | |
| | Total Bilirubin | | |
| | | umol/L | Pre-ECMO, t=12h, |
| | Amylase | iu/L | 24h, 48h, 72h ECMO |
| | CRP | mg/L | and 24h post ECMO |
| | Haemoglobin | g/L | and discharge |
| | Haematocrit | L/L | |
| | Platelet count | x10^9/L | |
| | INR | | |
| | APTT ratio | | |
| | Fibrinogen | g/L | |

| Туре | Variable | Unit/Reference | Time points |
|---|---|---|---|
| Outcome | Total hours on ECMO | hours | |
| | Alive at discharge | Y/N | |
| | Died | Y/N | |
| | Chest open | Y/N | |
| | Patient weaned from ECMO? | Y/N | |
| | Reintubation | Y/N | |
| | Fluid balance | ml | 12h, 24hr |
| | Bleeding cannulation site Urine output | ml | 12h, 24hr |
| | Any RBC transfused? | Y/N | Pre, during & post |
| | Any non RBC transfused? | y/N | ECMO |
| | Blood products transfused | ,<br>No of units | |
| | Volume transfused | ml | |
| | ICU length of stay | days | |
| | Hospital length of stay | days | |
| | ltem | | Score |
| Questionnaire | The fact that your baby's treatmen | nt involves research | 1 - 5 |
| • | What the researchers are trying to | | 1 - 5 |
| | How long your baby will be in the | 1 - 5 | |
| | The procedures your baby will und | · | 1 - 5 |
| | The possible disadvantages of part | • | 1 - 5 |
| | How participation in this study ma | , • | 1 - 5 |
| | The effect of the study on the con | 1 3 | |
| | records | indentiality of your baby silledical | 1 - 5 |
| | Whom you should contact if you h the study | ave questions or concerns about | 1 - 5 |
| | The fact that participation in the s | tudy is voluntary | 1 - 5 |
| | The fact that you can withdraw yo | ur baby from the study any moment | 1 - 5 |
| | Overall, how well did you understa consent form? | and the study when you signed the | 1 - 5 |